CLINICAL TRIAL: NCT01121718
Title: Real-Time NIR-Guided Sentinel Lymph Node Mapping in Melanoma
Brief Title: NIR-Guided Sentinel Lymph Node Mapping in Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Yolonda L. Colson, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-039
Record Dates: First submitted 2010-05-06; First posted 2010-05-12 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Melanoma
Keywords: lymph node
MeSH Terms: conditions — Melanoma | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: This is an experimental study. All study subjects will receive the same intervention.
Masking Description: This study does not involve any masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICG Intervention (Experimental): Intraoperative NIR fluorescence imaging was performed after injection of 1.0 ml of 100 µM, 250 µM or 500 µM of ICG:HSA in four quadrants around the primary lesion. (The intervention to be administered is the ICG.)
  Interventions: Drug: ICG Intervention

INTERVENTIONS:
Drug: ICG Intervention — NIR-guided sentinel lymph node mapping with indocyanine green (ICG)
  Other Names: NIR fluorescence imaging; Sentinel Lymph Node

SUMMARY:
This study will try to define an appropriate dose of the investigational drug indocyanine green (ICG) in combination with near infrared (NIR) imaging to use for future studies.

ICG is a dye which has been in use since the 50s, and is approved for testing liver function and measuring blood flow from the heart. It has been used in studies to map lymphatic pathways in lung and breast cancer and information from those studies suggest it may help identify lymph nodes associated with melanoma. ICG can be detected within the body using near-infrared light cameras.

In this study the investigators are looking at how easily ICG can get to the first lymph node (sentinel lymph node [SLN]) associated with melanoma, whether the investigators can see the path of the ICG and the SLN using a near infrared camera, and what dose of ICG works the best. While the current method for SNL mapping, known as lymphoscintigraphy, is effective it does provide a small amount of radiation. This study will compare the investigators results to the standard procedure.

DETAILED DESCRIPTION:
At the time of surgery, you will undergo a lymphoscintigraphic procedure which is standard of care for patients with melanoma. You will also receive a dose of ICG mixed with human serum albumin. This will be administered in four small injections immediately around your tumor or the tumor scar if it has already been removed. Pictures of the ICG solution will be taken with the NIR camera and the progression of the dye along the lymphatic channel from your tumor to the SLN will be monitored.

As each lymph node is removed, pictures will be taken to see if the ICG dye has entered and colored that node. We will compare this technique with the results from the lymphoscintigraphy to measure accuracy.

Patients will be followed for at least one hour post injection for adverse events. The patient will then be taken off of the study. The results from each intervention will subsequently analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma and an appropriate surgical candidate for a sentinel lymph node biopsy
* Stage of disease conducive to sentinel lymph node biopsy as determined by oncologic surgeon
* Receiving a planned lymphoscintigraphy procedure

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to indocyanine green, including those patients with a history of iodide or seafood allergy
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Feasibility | We will analyze data immediately following each case, and analyze all collected data at 6 month intervals
  To determine the feasibility of real-time intraoperative NIR lymphatic mapping with concurrent identification of the sentinel lymph node in human melanoma using indocyanine green.

SECONDARY OUTCOMES:
Comparison of SLN identification rate between near-infrared mapping and lymphoscintigraphy. | We will analyze data immediately following each case, and analyze all collected data at 6 month intervals

CONTACTS AND LOCATIONS:
Overall Officials: Yolonda Colson, MD, PhD, Principal Investigator — Dana Faber Cancer Institute / Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided
At this time, a plan is not in place to make IPD available to other researchers.